CLINICAL TRIAL: NCT02259595
Title: Randomized, Placebo-controlled, Double-blind, Dose Escalation Study to Determine the Safety, Tolerability, and Pharmacokinetic Profile of HPN-07 and HPN-07 Plus NAC in Single Doses in Male and Female Subjects
Brief Title: Study to Determine the Safety, Tolerability, and Pharmacokinetic Profile of HPN-07 and HPN-07 Plus NAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otologic Pharmaceutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPN-07-PK-101
Record Dates: First submitted 2014-09-02; First posted 2014-10-08 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Hearing Loss; Sensorineural Hearing Loss; Noise-Induced Hearing Loss
Keywords: Hearing Loss; Sensorineural Hearing Loss; Noise-Induced Hearing Loss; Antioxidant; NAC; N-acetylcysteine; HPN-07
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural; Hearing Loss, Noise-Induced | interventions — disufenton sodium; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HPN-07 500 mg / Placebo (Experimental): Single dose of 500mg HPN-07 plus placebo in oral capsules.
  Interventions: Drug: HPN-07; Drug: Placebo
- HPN-07 1000 mg / Placebo (Experimental): Single dose of 1,000mg HPN-07 plus placebo in oral capsules
  Interventions: Drug: HPN-07; Drug: Placebo
- HPN-07 1500 mg / Placebo (Experimental): Single dose of 1,500mg HPN-07 plus placebo in oral capsules
  Interventions: Drug: HPN-07; Drug: Placebo
- HPN-07 MTD plus NAC 1200mg (Experimental): Single dose of maximum tolerated dose of HPN-07 plus 1,200 mg NAC in oral capsules. Dose selection will be determined from safety data of previous cohorts by Data Assessment Committee (DAC).
  Interventions: Drug: HPN-07; Drug: NAC

INTERVENTIONS:
Drug: HPN-07 — 500-1,500 mg oral capsules administered in a single dose
  Other Names: disufenton sodium; Disodium 4-[(tert-butylimino)methyl]benzene-1,3-disulfonate N-oxide
Drug: NAC — 1,200mg NAC administered via oral capsule in single dose
  Other Names: N-acetylcysteine; acetylcysteine; N-acetyl-L-cysteine
  Arms: HPN-07 MTD plus NAC 1200mg
Drug: Placebo — placebo oral capsule
  Arms: HPN-07 1000 mg / Placebo; HPN-07 1500 mg / Placebo; HPN-07 500 mg / Placebo

SUMMARY:
This study is a single-center, randomized, placebo-controlled, double-blind, single ascending dose escalation study to determine the safety, tolerability, and PK profile of oral administration of HPN-07 in single doses to approximately 32 healthy male and female subjects between 18 and 55 years of age.

Subjects will receive single oral doses of the study drug. The primary endpoint of this trial is to establish the safety and tolerability of HPN-07 and HPN-07 plus N-acetylcysteine (NAC).

DETAILED DESCRIPTION:
This study is a single-center, randomized, placebo-controlled, double-blind, single ascending dose escalation study to determine the safety, tolerability, and PK profile of oral administration of HPN-07 in single doses to healthy male and female subjects between 18 and 55 years of age.

Approximately 32 subjects will be enrolled in a panel of 4 cohorts with approximately 8 subjects per cohort. There will be approximately 3 sequential ascending dosing levels of HPN-07, with each cohort administered 1 dose of HPN-07 ranging from 500 mg to 1,500 mg and the fourth cohort administered the highest tolerated dose of HPN-07 plus 1,200 mg NAC.

The primary endpoint of this trial is to establish the safety and tolerability of HPN-07 and HPN-07 plus N-acetylcysteine (NAC). Pharmacokinetics (PK) analysis of HPN-07 will enable a preliminary determination of the relationship between dose and the time course of the drug concentration in the body. Blood samples will be collected at regular intervals over the predicted time of HPN-07 systemic exposure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18-55 years of age (inclusive), at the time of enrollment.
* Healthy as judged by a responsible physician with no clinically significant abnormality identified on the medical or laboratory evaluation, including 12-lead electrocardiogram (ECG). A subject with a clinical abnormality or laboratory parameters outside the reference range for this age group may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures (as defined as the research site's standard operating procedures).
* Male subjects who are surgically sterile OR agree to abstain from sexual intercourse with a female partner OR agree to use a condom and spermicide during sexual intercourse with a female partner who meets the following criteria: 1) uses another form of contraception, such as an intrauterine device (IUD), occlusive cap (diaphragm or cervical/vault cap) with spermicide, oral contraceptives, injectable progesterone, subdermal implants, female condom, contraceptive patch, or contraceptive vaginal ring; and/or 2) has had a tubal ligation or hysterectomy. These criteria must be followed from the time of the first dose of study medication until 14 days after the last dose of study medication. Men must also abstain from sperm donation from the time of the first dose of study medication until 14 days after the last dose of study medication.
* Female subjects of childbearing potential must be practicing abstinence or are using, and willing to continue using, a medically acceptable form of birth control for at least 1 month prior to Screening (at least 3 months for hormonal contraceptives) and for at least 2 months after the last study drug administration. Medically acceptable forms of contraception include abstinence, hormonal contraceptives (oral, patch or vaginal ring), intrauterine device, progestin implant or injection, bilateral tubal ligation, or double-barrier methods (i.e., male condom in addition to a diaphragm or a contraceptive sponge).
* Female subjects of non-childbearing potential, defined as: having undergone successful surgical sterilization (hysterectomy and/or bilateral oophorectomy/salpingo-oophorectomy, as determined by subject medical history) or post-menopausal. Postmenopausal is defined as being amenorrheic for at least 1 year without another cause and a follicle-stimulating hormone (FSH) level ~50 mlU/ml.
* Female subjects must have a negative pregnancy test at screening and Day -1 (admission).
* Minimum body weight of 50.0 kg and body mass index (BMI) between 18.0 kg/m2 and 33.0 kg/m2 (inclusive).
* Non-smoker (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc:, for 6 months prior to the administration of the study medication) and has negative findings on a breath carbon monoxide (CO) test.
* Willing and able to comply with study instructions and commit to all follow-up visits, and willing and able to abide by all study requirements and restrictions.
* Ability to understand, agree to, and sign the study informed consent form (ICF) prior to initiation of any protocol related procedures.

Exclusion Criteria:

* Self-reported substance or alcohol dependence or abuse (excluding nicotine and caffeine) within the past 2 years, as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and/or subjects who have ever been in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence.
* History of serious adverse reactions or hypersensitivity to any drug; or known allergy to any of the test product(s), or any components in the test product(s); or history of hypersensitivity; or allergic reactions to any of the study preparations as described in the Investigator's Brochure; or severe allergic reaction (including anaphylaxis) to any food, or bee stings or previous status asthmaticus.
* History of renal stones or taking cardiac nitrates.
* Any clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator, may place the subject at an unacceptable risk as a participant in this trial or may interfere with the distribution, metabolism, or excretion of drugs.
* Abnormal physical findings of clinical significance, at screening or on Day -1, which would interfere with the objectives of the study.
* History or presence of orthostatic hypotension (~20 mmHg drop in systolic blood pressure, or ~10 mmHg drop in diastolic blood pressure, or subject experiences lightheadedness or dizziness) at screening or on Day-1.
* Clinically significant abnormal laboratory values (as determined by the Investigator) at the screening evaluation.
* Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
* 12-lead ECG obtained at screening with PR >240 msec, QRS >110 msec, and QTc >440 msec for males and >450 msec for females, bradycardia (<50 bpm), or clinically significant minor ST wave changes on the screening ECG or any other changes on the screening ECG that would interfere with measurement of the QT interval.
* Major surgical interventions within 6 months before the study.
* Has a positive pre-study hepatitis B surface antigen; positive hepatitis C virus (HCV) antibody or detectable HCV ribonucleic acid (RNA); or positive human immunodeficiency virus (HIV) antibody result.
* Use of a prohibited medication or supplement, as specified in Section 9.6.
* Has a history of regular alcohol consumption averaging >14 drinks/week for men and >9 drinks/week for women (1 drink (10 g alcohol] = 100 ml of wine or 280 ml of standard strength beer or 30 ml of 80 proof distilled spirits) within 6 months of the screening visit.
* Loss of 500 ml, or more, of blood during the 3-month period before the drug administration, e.g., blood donor.
* Symptoms of a significant somatic or mental illness in the 4-week period preceding drug administration, as per investigator discretion.
* Exclude subjects with a positive breath alcohol test or urine drug screen at screening. Suspected false positive results may be repeated at the discretion of the Investigator.
* Concurrent participation in another drug or device research study or within 30 days of participation in another drug or device research study.
* Considered by the Investigator to be an unsuitable candidate for this study.
* Women who are breastfeeding, pregnant, or intend to become pregnant during the course of the study.
* An employee of the sponsor or research site personnel directly affiliated with this study or their immediate family members defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single doses of HPN-07, alone and in co-administration with NAC: Adverse events | 48 hours
  The primary endpoint of this trial is to establish the safety and tolerability of HPN-07 and HPN-07 plus NAC. The following safety parameters will be evaluated for adverse events as determined by: 12-lead ECG, clinical laboratory tests, urinalysis, and vital signs.

SECONDARY OUTCOMES:
Area under the curve (AUC) of single doses of HPN-07, alone and in co-administration with NAC | pre-dose, 5, 15, and 30 min, and 1, 2, 4, 6, 8, 12, 24, and 48h post dosing
Maximum observed plasma concentration (Cmax) of single doses of HPN-07, alone and in co-administration with NAC | pre-dose, 5, 15, and 30 min, and 1, 2, 4, 6, 8, 12, 24, and 48h post dosing
Half life (t1/2) of single doses of HPN-07, alone and in co-administration with NAC | pre-dose, 5, 15, and 30 min, and 1, 2, 4, 6, 8, 12, 24, and 48h post dosing
Volume of distribution (Vz) of single doses of HPN-07, alone and in co-administration with NAC | pre-dose, 5, 15, and 30 min, and 1, 2, 4, 6, 8, 12, 24, and 48h post dosing
Mean transit time (MTT) of single doses of HPN-07, alone and in co-administration with NAC | pre-dose, 5, 15, and 30 min, and 1, 2, 4, 6, 8, 12, 24, and 48h post dosing
Total clearance (CL) of single doses of HPN-07, alone and in co-administration with NAC | pre-dose, 5, 15, and 30 min, and 1, 2, 4, 6, 8, 12, 24, and 48h post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Treva Tyson, MD, Principal Investigator — Wake Research Associates
Locations (1):
- Wake Research Associates, Raleigh, North Carolina, United States